CLINICAL TRIAL: NCT02651857
Title: Exploratory Study of Upper and Lower Endoscopic Fuse System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EndoChoice Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Exploratory study
Record Dates: First submitted 2016-01-05; First posted 2016-01-11 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2016-01

CONDITIONS: Gastrointestinal Diseases
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endoscopy exploratory single arm (Experimental)
  Interventions: Device: Fuse® Colonoscope; Device: Fuse® Gastroscope

INTERVENTIONS:
Device: Fuse® Colonoscope — Endoscopic diagnostic procedures for lower GI tract
Device: Fuse® Gastroscope — Endoscopic diagnostic procedures for upper GI tract

SUMMARY:
Single-Center, Exploratory Study of EndoChoice's Upper and Lower Gastrointestinal Endoscopic Systems Utilizing EndoChoice's Full Spectrum Optical Technology

DETAILED DESCRIPTION:
The investigational devices are EndoChoice gastrointestinal endoscopic systems that are similar in their fit, form, and functions to the corresponding commercially available models with the exception of the EndoChoice's proprietary Optical system that enhances their field of view.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients ages of 18-75
* The patient has been scheduled for routine screening upper or lower endoscopy, diagnostic endoscopic work up, or endoscopic surveillance.
* Signed informed consent form

Exclusion Criteria:

* Patients who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the patient's participation in this study.
* Patients who are unable to consent
* Pregnant female patients of any age.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27

PRIMARY OUTCOMES:
Performance, usability and ease of use (performance questionnaire) | Through study completion, estimate average of 1 year
  The performance of the device is assessed via a performance questionnaire which the recruiting (and treatment providing) physician will answer

SECONDARY OUTCOMES:
Safety (adverse and severe adverse events) | Through study completion, estimate average of 1 year
  Establish safety of the device by measure of adverse and severe adverse events, if such occur.

IPD SHARING:
Plan to Share IPD: Undecided